CLINICAL TRIAL: NCT01124045
Title: A Phase IIIB, Multicenter, Randomized, Double-Masked, Parallel-Group, Active-Controlled Study of the Safety and Efficacy of Difluprednate Ophthalmic Emulsion, 0.05% (Durezol™) 4 Times Daily (QID) and Prednisolone Acetate Ophthalmic Suspension, 1.0% (Pred Forte™) QID for the Treatment of Inflammation Following Cataract Surgery in Children 0 to 3 Years of Age
Brief Title: Difluprednate Pediatric Study for the Treatment of Inflammation Post-Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-10-004
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-04

CONDITIONS: Cataracts; Inflammation
Keywords: Pediatric; Cataracts; Inflammation; Durezol; Pred Forte; Difluprednate; Prednisolone
MeSH Terms: conditions — Cataract; Inflammation | interventions — difluprednate; prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DUREZOL (Experimental): Difluprednate ophthalmic emulsion, 0.05%, 1 drop in the study eye at the end of surgery (Day 0) and 4 times a day beginning on the day after surgery (Day 1) for 14 days, followed by a tapering period of 14 days, dependent upon the Investigator's determination of adequate response to treatment
  Interventions: Drug: Difluprednate ophthalmic emulsion, 0.05%
- PRED FORTE (Active Comparator): Prednisolone acetate ophthalmic suspension, 1.0%, 1 drop in the study eye at the end of surgery (Day 0) and 4 times a day beginning on the day after surgery (Day 1) for 14 days, followed by a tapering period of 14 days, dependent upon the Investigator's determination of adequate response to treatment
  Interventions: Drug: Prednisolone acetate ophthalmic suspension, 1.0%

INTERVENTIONS:
Drug: Difluprednate ophthalmic emulsion, 0.05% — Topical ocular administration
  Other Names: DUREZOL™
  Arms: DUREZOL
Drug: Prednisolone acetate ophthalmic suspension, 1.0% — Topical ocular administration
  Other Names: PRED FORTE™
  Arms: PRED FORTE

SUMMARY:
The primary objective of this study was to compare the safety and efficacy of Durezol™ compared to Pred Forte™ for the treatment of inflammation following cataract surgery in a pediatric population 0 to 3 years of age.

DETAILED DESCRIPTION:
Parents or guardians instilled patients' assigned study medications once on the day of surgery (Day 0) and 4 times daily (QID) beginning on the day after surgery (Day 1) for 14 days followed by a tapering period of 14 days (dependent upon the Investigator's determination of adequate response to treatment). Patients were evaluated for safety and efficacy on the following visits: Day 0 (day of surgery), Day 1, Day 8 ± 1 day, Day 15 ± 2 days and Day 29 ± 2 days (end of study drug treatment). Additional safety visits occurred at 1 week after the last dose + 2 days and at 3 Months + 1 week. No inferential statistical analysis was planned for this study. Data was summarized using descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 3 years of age.
* Undergoing uncomplicated cataract extraction in 1 eye with or without intraocular lens.
* Informed consent signed by a parent or legal guardian.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Presence of any active or suspected viral, bacterial, or fungal disease in the study eye.
* Use of any topical medication in the study within 7 days prior to surgery, except for drops that are needed to examine the eye or to prepare for surgery.
* Patients with posttraumatic cataract.
* Active uveitis in the study eye.
* Ocular neoplasm in the study eye.
* Human immunodeficiency virus (HIV); acquired immunodeficiency syndrome (AIDS).
* Suspected permanent low vision or blindness in the fellow nonstudy eye. The study eye must not be the patient's only good eye.
* Patients on systemic steroids or nonsteroidal anti-inflammatory drugs.
* History of steroid-induced intraocular pressure (IOP) rise.
* Currently on medication for ocular hypertension or glaucoma in the study eye.
* Diabetes.
* Other protocol-defined exclusion criteria may apply.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and recruited from 17 study centers located within the United States.
Pre-assignment Details: This reporting group includes all patients who were exposed to the study drug. One patient randomized to DUREZOL withdrew consent prior to receiving study medication.
Period: Overall Study
Arm/Group | DUREZOL | PRED FORTE
Started | 39 | 40
Completed | 39 | 37
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all patients who were exposed to the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | DUREZOL | PRED FORTE | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Customized [Number; unit: participants]
  Newborns: 0 to 27 days | 3 | 3 | 6
  Infants and Toddlers: 28 days to 23 months | 28 | 26 | 54
  Children: 2 to 3 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With an Anterior Cell Grade of 0 (no Cells) at Day 15 ± 2 Days
Description: Anterior cell grade was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 5-point scale: Grade 0=0 cells; Grade 1=1 to 10 cells; Grade 2=11 to 20 cells; Grade 3=21 to 50 cells; Grade 4=>50 cells. The presence of blood cells (red and white) in the anterior chamber of the eye (the fluid-filled space inside the eye between the iris and the cornea's innermost surface) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation.
Time Frame: Day 15 ± 2 days
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication. One patient (DUREZOL) had missing anterior cell grade assessment at all visits.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 38 | 40
Percentage of patients | 78.9 | 77.5

2. Secondary Outcome: Global Assessment Score of Postoperative Inflammation by Visit
Description: A Global Assessment Score (GAS) was assigned by the Investigator based on the clinical evidence of postoperative inflammation: 0=clear, 1=improving satisfactorily; 2=not improving or worsening, withdrawal from study indicated to allow appropriate alternative therapy to be instituted. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 30.8 | 17.5
  Day 1: Grade 1 | 69.2 | 82.5
  Day 1: Grade 2 | 0.0 | 0.0
  Day 8: Grade 0 | 48.7 | 25.0
  Day 8: Grade 1 | 48.7 | 70.0
  Day 8: Grade 2 | 2.6 | 5.0
  Day 15: Grade 0 | 56.4 | 50.0
  Day 15: Grade 1 | 43.6 | 50.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 29: Grade 0 | 79.5 | 72.5
  Day 29: Grade 1 | 20.5 | 25.0
  Day 29: Grade 2 | 0.0 | 2.5
  1 Week after Last Dose: Grade 0 | 89.7 | 90.0
  1 Week after Last Dose: Grade 1 | 7.7 | 7.5
  1 Week after Last Dose: Grade 2 | 2.6 | 2.5
  Month 3: Grade 0 | 92.3 | 92.5
  Month 3: Grade 1 | 5.1 | 7.5
  Month 3: Grade 2 | 2.6 | 0.0

3. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Anterior Chamber Cell Grade
Description: Anterior chamber cell grade was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 5-point scale: Grade 0=0 cells; Grade 1=1 to 10 cells; Grade 2=11 to 20 cells; Grade 3=21 to 50 cells; Grade 4=>50 cells. The presence of blood cells (red and white) in the anterior chamber of the eye (the fluid-filled space inside the eye between the iris and the cornea's innermost surface) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication. One patient had missing anterior cell grade assessment at all visits.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 38 | 40
Percentage of patients
  Day 1: Grade 0 | 23.7 | 40.0
  Day 1: Grade 1 | 57.9 | 30.0
  Day 1: Grade 2 | 15.8 | 27.5
  Day 1: Grade 3 | 2.6 | 0.0
  Day 1: Grade 4 | 0.0 | 2.5
  Day 8: Grade 0 | 55.3 | 57.5
  Day 8: Grade 1 | 36.8 | 32.5
  Day 8: Grade 2 | 5.3 | 10.0
  Day 8: Grade 3 | 2.6 | 0.0
  Day 8: Grade 4 | 0.0 | 0.0
  Day 15: Grade 0 | 78.9 | 77.5
  Day 15: Grade 1 | 18.4 | 17.5
  Day 15: Grade 2 | 0.0 | 5.0
  Day 15: Grade 3 | 2.6 | 0.0
  Day 15: Grade 4 | 0.0 | 0.0
  Day 29: Grade 0 | 89.5 | 95.0
  Day 29: Grade 1 | 10.5 | 2.5
  Day 29: Grade 2 | 0.0 | 2.5
  Day 29: Grade 3 | 0.0 | 0.0
  Day 29: Grade 4 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 97.4 | 95.0
  1 Week after Last Dose: Grade 1 | 2.6 | 2.5
  1 Week after Last Dose: Grade 2 | 0.0 | 2.5
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  1 Week After Last Dose: Grade 4 | 0.0 | 0.0
  Month 3: Grade 0 | 94.7 | 97.5
  Month 3: Grade 1 | 5.3 | 0.0
  Month 3: Grade 2 | 0.0 | 2.5
  Month 3: Grade 3 | 0.0 | 0.0
  Month 3: Grade 4 | 0.0 | 0.0

4. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Anterior Chamber Flare Grade
Description: Anterior chamber flare was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. The presence of flare (increased protein levels) in the anterior chamber of the eye (the fluid-filled space inside the eye between the iris and the cornea's innermost surface) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 38 | 40
Percentage of patients
  Day 1: Grade 0 | 41.0 | 45.0
  Day 1: Grade 1 | 51.3 | 37.5
  Day 1: Grade 2 | 7.7 | 12.5
  Day 1: Grade 3 | 0.0 | 5.0
  Day 8: Grade 0 | 61.5 | 52.5
  Day 8: Grade 1 | 35.9 | 40.0
  Day 8: Grade 2 | 2.6 | 5.0
  Day 8: Grade 3 | 0.0 | 2.5
  Day 15: Grade 0 | 74.4 | 70.0
  Day 15: Grade 1 | 17.9 | 27.5
  Day 15: Grade 2 | 7.7 | 2.5
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 87.2 | 92.5
  Day 29: Grade 1 | 12.8 | 7.5
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 94.9 | 92.5
  1 Week after Last Dose: Grade 1 | 2.6 | 7.5
  1 Week after Last Dose: Grade 2 | 2.6 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 92.3 | 95.0
  Month 3: Grade 1 | 5.1 | 5.0
  Month 3: Grade 2 | 2.6 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

5. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Corneal Clarity
Description: Corneal clarity was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Lack of corneal clarity (1-3) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 92.3 | 87.5
  Day 1: Grade 1 | 7.7 | 12.5
  Day 1: Grade 2 | 0.0 | 0.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 94.9 | 90.0
  Day 8: Grade 1 | 5.1 | 7.5
  Day 8: Grade 2 | 0.0 | 2.5
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 94.9 | 90.0
  Day 15: Grade 1 | 5.1 | 10.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 97.4 | 97.5
  Day 29: Grade 1 | 2.6 | 2.5
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 97.5
  1 Week after Last Dose: Grade 1 | 0.0 | 2.5
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 97.5
  Month 3: Grade 1 | 0.0 | 2.5
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

6. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Conjunctival Injection
Description: Conjunctival injection was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Conjunctival injection (redness of the white sclera of the eye) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 46.2 | 25.0
  Day 1: Grade 1 | 48.7 | 65.0
  Day 1: Grade 2 | 2.6 | 10.0
  Day 1: Grade 3 | 2.6 | 0.0
  Day 8: Grade 0 | 79.5 | 77.5
  Day 8: Grade 1 | 20.5 | 22.5
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 89.7 | 92.5
  Day 15: Grade 1 | 10.3 | 7.5
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 97.4 | 95.0
  Day 29: Grade 1 | 2.6 | 5.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

7. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Ciliary/Limbal Injection
Description: Ciliary/limbal injection was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Ciliary/limbal injection (redness of the white sclera of the eye near the limbal ring) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 69.2 | 57.5
  Day 1: Grade 1 | 28.2 | 40.0
  Day 1: Grade 2 | 0.0 | 2.5
  Day 1: Grade 3 | 2.6 | 0.0
  Day 8: Grade 0 | 89.7 | 90.0
  Day 8: Grade 1 | 10.3 | 10.0
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 100.0
  Day 15: Grade 1 | 0.0 | 0.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 97.5
  Day 29: Grade 1 | 0.0 | 2.5
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

8. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Chemosis
Description: Chemosis was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Chemosis (swelling of the conjunctiva) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 82.1 | 85.0
  Day 1: Grade 1 | 15.4 | 15.0
  Day 1: Grade 2 | 0.0 | 0.0
  Day 1: Grade 3 | 2.6 | 0.0
  Day 8: Grade 0 | 97.4 | 100.0
  Day 8: Grade 1 | 2.6 | 0.0
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 97.5
  Day 15: Grade 1 | 0.0 | 2.5
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 100.0
  Day 29: Grade 1 | 0.0 | 0.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

9. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Hypopyon
Description: Hypopyon was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Hypopyon (pus in the anterior chamber of the eye) is a sign of ocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 100.0 | 100.0
  Day 1: Grade 1 | 0.0 | 0.0
  Day 1: Grade 2 | 0.0 | 0.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 100.0 | 100.0
  Day 8: Grade 1 | 0.0 | 0.0
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 100.0
  Day 15: Grade 1 | 0.0 | 0.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 100.0
  Day 29: Grade 1 | 0.0 | 0.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

10. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Vitritis
Description: Vitritis was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Vitritis (accumulation of inflammatory cells or exudates in the vitreous humor, the fluid that fills the middle chamber of the eye) is a sign of ocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 100.0 | 97.5
  Day 1: Grade 1 | 0.0 | 2.5
  Day 1: Grade 2 | 0.0 | 0.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 100.0 | 97.5
  Day 8: Grade 1 | 0.0 | 0.0
  Day 8: Grade 2 | 0.0 | 2.5
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 97.5
  Day 15: Grade 1 | 0.0 | 0.0
  Day 15: Grade 2 | 0.0 | 2.5
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 97.5
  Day 29: Grade 1 | 0.0 | 0.0
  Day 29: Grade 2 | 0.0 | 2.5
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 97.5
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 2.5
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 97.5
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 2.5
  Month 3: Grade 3 | 0.0 | 0.0

11. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Wound Integrity
Description: Wound integrity was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Lack of wound integrity (healing, 1-3) is a sign of inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 100.0 | 100.0
  Day 1: Grade 1 | 0.0 | 0.0
  Day 1: Grade 2 | 0.0 | 0.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 100.0 | 100.0
  Day 8: Grade 1 | 0.0 | 0.0
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 100.0
  Day 15: Grade 1 | 0.0 | 0.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 100.0
  Day 29: Grade 1 | 0.0 | 0.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 1: Grade 0 | 100.0 | 100.0
  Month 1: Grade 1 | 0.0 | 0.0
  Month 1: Grade 2 | 0.0 | 0.0
  Month 1: Grade 3 | 0.0 | 0.0

12. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Photophobia
Description: Photophobia was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Photophobia (abnormal intolerance to visual perception of light) is a symptom of intraocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 71.8 | 60.0
  Day 1: Grade 1 | 20.5 | 35.0
  Day 1: Grade 2 | 7.7 | 5.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 89.7 | 87.5
  Day 8: Grade 1 | 10.3 | 10.0
  Day 8: Grade 2 | 0.0 | 2.5
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 97.4 | 95.0
  Day 15: Grade 1 | 2.6 | 5.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 97.4 | 92.5
  Day 29: Grade 1 | 2.6 | 5.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 2.5
  1 Week after Last Dose: Grade 0 | 100.0 | 97.5
  1 Week after Last Dose: Grade 1 | 0.0 | 2.5
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

13. Secondary Outcome: Global Assessment of Inflammation - Individual Component Scoring by Visit: Lacrimation
Description: Lacrimation was assessed by the Investigator during slit lamp or ophthalmoscopy/light examination and graded on a 4-point scale: 0=absent; 1=mild; 2=moderate; 3=severe. Excessive lacrimation (tear production and secretion, 1-3) is a symptom of ocular inflammation. A score of 0 indicates an absence of inflammation. For this outcome measure, percentage of patients by grade and visit is reported.
Time Frame: Day 1, Day 8 ± 1 day, Day 15 ± 2 days, Day 29 ± 2 days, 1 Week after Last Dose + 2 days, 3 Months + 1 week
Population: Intent-to-treat (ITT): All patients who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of patients
Arm/Group | DUREZOL | PRED FORTE
Number analyzed (Participants) | 39 | 40
Percentage of patients
  Day 1: Grade 0 | 64.1 | 72.5
  Day 1: Grade 1 | 30.8 | 22.5
  Day 1: Grade 2 | 5.1 | 5.0
  Day 1: Grade 3 | 0.0 | 0.0
  Day 8: Grade 0 | 94.9 | 97.5
  Day 8: Grade 1 | 5.1 | 2.5
  Day 8: Grade 2 | 0.0 | 0.0
  Day 8: Grade 3 | 0.0 | 0.0
  Day 15: Grade 0 | 100.0 | 95.0
  Day 15: Grade 1 | 0.0 | 5.0
  Day 15: Grade 2 | 0.0 | 0.0
  Day 15: Grade 3 | 0.0 | 0.0
  Day 29: Grade 0 | 100.0 | 100.0
  Day 29: Grade 1 | 0.0 | 0.0
  Day 29: Grade 2 | 0.0 | 0.0
  Day 29: Grade 3 | 0.0 | 0.0
  1 Week after Last Dose: Grade 0 | 100.0 | 100.0
  1 Week after Last Dose: Grade 1 | 0.0 | 0.0
  1 Week after Last Dose: Grade 2 | 0.0 | 0.0
  1 Week after Last Dose: Grade 3 | 0.0 | 0.0
  Month 3: Grade 0 | 100.0 | 100.0
  Month 3: Grade 1 | 0.0 | 0.0
  Month 3: Grade 2 | 0.0 | 0.0
  Month 3: Grade 3 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. The safety population includes all patients who were exposed to the study drug.
Description: An adverse event was considered to be any untoward medical occurrence in the health of a patient who was exposed to study medication, regardless of causal relationship with the study medication. Adverse events were obtained as solicited comments from the study patients and as observations by the study Investigator as outlined in the study protocol.
Arm/Group | DUREZOL | PRED FORTE
Serious Adverse Events (participants affected / at risk) | 8/39 | 11/40
Other Adverse Events (participants affected / at risk) | 16/39 | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DUREZOL (N=39) | PRED FORTE (N=40)
Medical observation (Investigations) | 6 | 10 — Not related. Hospital admission was required for procedures involving surgery/anesthesia of certain infants.
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 — Not related
Intraocular pressure increased (Investigations) | 1 | 0 — Related
Cataract cortical (Immune system disorders) | 1 | 0 — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DUREZOL (N=39) | PRED FORTE (N=40)
Conjunctivitis (Eye disorders) | 3 | 0
Posterior capsule opacification (Eye disorders) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 2
Ear infection (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 0
Intraocular pressure increased (Investigations) | 2 | 1
Cataract operation (non-study eye) (Surgical and medical procedures) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.